CLINICAL TRIAL: NCT02467387
Title: A Phase IIa Randomized Study to Assess the Safety, Tolerability, and Preliminary Efficacy of a Single Intravenous Dose of Ischemia-tolerant Allogeneic Mesenchymal Bone Marrow Cells to Subjects With Non-ischemic Heart Failure
Brief Title: A Study to Assess the Effect of Intravenous Dose of (aMBMC) to Subjects With Non-ischemic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CardioCell LLC (Industry)
Collaborators: Stemedica Cell Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STEM-104-M-CHF; NCT02123706 (obsolete NCT alias)
Record Dates: First submitted 2015-06-02; First posted 2015-06-10 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Non-Ischemic Heart Failure
Keywords: Non-ischemic Heart Failure; Stem Cells
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Human (aMBMC) (Experimental): Intervention: One time intravenous infusion of 1.5 million (aMBMC) per kg administered at approximately 2mL/min. Maximum dose as for 100kg subject or 150 million cells for any subject 100kg or more.
  Interventions: Drug: Allogeneic Mesenchymal Bone Marrow Cells (aMBMC)
- Placebo:Lactated Ringer's Solution (LRS) (Placebo Comparator): Intervention: One time intravenous infusion of 1.5mL/kg Lactated Ringer's Solution (LRS) administered at a constant rate of approximately 2mL/min.
  Interventions: Drug: Lactated Ringer's Solution

INTERVENTIONS:
Drug: Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) — One time infusion Allogeneic Mesenchymal Bone Marrow Cells (aMBMC) 1.5 million cells/kg.
  Other Names: Mesenchymal Stem Cells, (MSC) Marrow Stromal Cells.
  Arms: Experimental: Human (aMBMC)
Drug: Lactated Ringer's Solution — One time infusion 1.5mL/kg
  Other Names: (LRS)
  Arms: Placebo:Lactated Ringer's Solution (LRS)

SUMMARY:
A phase IIa study to assess the safety and preliminary efficacy of intravenous dose of ischemia-tolerant Allogeneic Mesenchymal Bone Marrow Cells in subjects with non-ischemic heart failure.

DETAILED DESCRIPTION:
A phase IIa, single-blind, placebo-controlled, crossover, multi-center, randomized study to assess the safety, tolerability, and preliminary efficacy of a single intravenous dose of ischemia-tolerant allogeneic mesenchymal bone marrow cells to subjects with heart failure of non-ischemic etiology.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age
2. LVEF ≤35% on echocardiogram within 12 months of randomization to undergo MRI
3. Screening cardiac MRI at baseline with:

   Ejection fraction ≤40% No significant hyper enhancement on MRI scan in the opinion of the central imaging lab reviewer
4. Patients with non-ischemic heart failure etiology, as documented by absent or non-obstructive coronary artery disease on x-ray angiography or coronary computed tomography
5. Patients with history of heart failure and treated for at least three months with GDMT
6. NYHA class II-III symptoms
7. Ability to understand and provide signed informed consent
8. Reasonable expectation that patient will receive standard post-treatment care and attend all scheduled safety follow-up visits

Exclusion Criteria:

1. Pregnant or nursing women or those of childbearing age and not using an effective method of contraception
2. History of stroke within 3 months
3. Cardiac surgery within 3 months prior to randomization or the likelihood of a requirement for such procedures during the study period
4. Current ICD or CRT or implantation planned within 6 months of infusion
5. Presence of clinically significant, uncorrected valvular heart disease, hypertrophic or restrictive cardiomyopathy, active myocarditis, or uncontrolled hypertension
6. History of cardiac arrest or life-threatening arrhythmias within 3 months
7. Treatment with parenteral inotropic agents within 1 month of randomization
8. Anticipated cardiac transplantation within 1 year
9. Illness other than heart failure with life expectancy less than 1 year
10. Received an experimental drug or device within 30 days of randomization
11. Left ventricular assist device or implantation planned in the next 6 months
12. Patients with complex congenital heart disease
13. Uncontrolled seizure disorder
14. Presence of immune deficiency
15. Clinically significant hematologic, hepatic, or renal impairment as determined by screening clinical laboratory tests:

    * Liver disease = ALT or AST > 3x normal, alkaline phosphatase or bilirubin >2x normal)
    * Renal disease = estimated glomerular filtration rate as assessed by the MDRD formula <30 ml/min
    * Hematologic = Unexplained leukocytosis >10 or hemoglobin < 9gm/dl
16. Presence of any other clinically-significant medical condition, psychiatric condition, or laboratory abnormality, that in the judgment of the investigator or sponsor for which participation in the study would pose a safety risk to the subject
17. Inability to comply with the conditions of the protocol
18. Malignancy within the previous five years, except adequately treated basal cell carcinoma, provided that it is neither infiltrating nor sclerosing, and carcinoma in situ of the cervix
19. Active myocarditis or early postpartum cardiomyopathy (within six months).
20. Systemic corticosteroids, cytostatics, immunosuppressive drug therapy (cyclophosphamide, methotrexate, cyclosporine, azathioprine, etc.), and DNA depleting or cytotoxic drugs taken within four weeks prior to study treatment
21. Porphyria
22. Allergy to sodium citrate or any "caine" type of local anesthetic
23. Any contraindication for gadolinium use for MRI
24. Patient scheduled for hospice care
25. Clinically relevant abnormal findings in the clinical history, physical examination, ECG, or laboratory tests at the screening assessment that would interfere with the objectives of the study or would preclude safe completion of the study. Abnormal findings could include: known HIV infection or other immunodeficiency state, chronic active viral infection (such as hepatitis B or C), acute systemic infections (defined as patients undergoing treatment with antibiotics), gastrointestinal tract bleeding, or any severe or acute concomitant illness or injury
26. Any other medical, social, or geographical factor that would make it unlikely that the patient could comply with study procedures (e.g., alcohol abuse, lack of permanent residence, severe depression, disorientation, distant location, or noncompliance)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristrun Stardal, RN, BSN, Study Director — Clinical Operations Manager
Locations (5):
- United States (5):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern University Centers for Heart Failure Therapy, Chicago, Illinois
  - Stony Brook Heart Institute, Stony Brook, New York
  - Hospital of the University of Pennsylvania, Heart Failure and Transplant Program, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Butler J, Epstein SE, Greene SJ, Quyyumi AA, Sikora S, Kim RJ, Anderson AS, Wilcox JE, Tankovich NI, Lipinski MJ, Ko YA, Margulies KB, Cole RT, Skopicki HA, Gheorghiade M. Intravenous Allogeneic Mesenchymal Stem Cells for Nonischemic Cardiomyopathy: Safety and Efficacy Results of a Phase II-A Randomized Trial. Circ Res. 2017 Jan 20;120(2):332-340. doi: 10.1161/CIRCRESAHA.116.309717. Epub 2016 Nov 16. PMID 27856497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 patients have been screened for eligibility between June, 2014 and April, 2016 at Emory University Medical Center, Atlanta, GA, Northwestern University Medical Center, Chicago, IL, University of Pennsylvania Medical Center, Philadelphia, PA, and Stony Brook University Medical Center, Stony Brook, NY.
Pre-assignment Details: 23 out of 34 patients have been randomized and 22 received the study intervention. Of those not randomized, 10 did not meet inclusion criteria and 1 could not tolerate CMR.
Groups:
- itMSC, Then Placebo: Participants first received itMSC 1.5 million per kilogram of weight, infused in the corresponding hospital facility at speed of 1 mL/minute (cell concentration 1 million/mL). After 90 days patients completed treatment at 90 days, and thus constituted the control treatment. After 90 day follow-up testing patients received Placebo and followed up for another 90 days. Total efficacy follow-up - 180 days. Safety measurements 0, 60, 90, days 270 and 450.
- Placebo, Then itMSC: Participants first received Placebo, infused in the corresponding hospital facility at speed of 1 mL/minute. After 90 days patients completed Placebo Control and related testing, and received itMSC treatment 1.5 million per kilogram of weight, and thus constituted the itMSC treated group for another 90 days.Total efficacy follow-up - 180 days. Safety measurements 0, 60, 90, days 270 and 450.
Period: First Intervention
Arm/Group | itMSC, Then Placebo | Placebo, Then itMSC
Started | 11 | 12
Received Treatment as Randomized | 10 | 12
Completed | 10 | 12
Not Completed | 1 | 0
Period: Second Intervention
Arm/Group | itMSC, Then Placebo | Placebo, Then itMSC
Started | 10 | 12
Completed | 7 | 12
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Population: itMSC, then Placebo: Participants first received itMSC 1.5 million per kilogram of weight, infused in the corresponding hospital facility at speed of 1 mL/minute (cell concentration 1 million/mL). After 90 days patients completed treatment at 90 days, and thus constituted the control treatment. After 90 day follow-up testing patients received Placebo and followed up for another 90 days. Total efficacy follow-up - 180 days. Safety follow-up - 240 days.
  Placebo, then itMSC: Participants first received Placebo, infused in the corresponding hospital facility at speed of 1 mL/minute. After 90 days patients completed Placebo Control and related testing, and received itMSC treatment 1.5 million per kilogram of weight, and thus constituted the itMSC treated group for another 90 days.Total efficacy follow-up - 180 days. Safety follow-up - 240 days. and thus constituted the control treatment.
Arm/Group | Study Population
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 92.5 (19.96)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.24 (7.56)
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — NYHA Class:
  Class I (Mild): Patients with cardiac disease but without resulting in limitation of physical activity.
  Class II (Mild): Cardiac disease resulting in slight limitation of physical activity.
  Class III (Moderate): Cardiac disease resulting in marked limitation of physical activity.
  Class IV (Severe): Cardiac disease resulting in the inability to carry on any physical activity without discomfort.
  Improvement in NYHA classification was analyzed using logistic regression with treatment and group assignment (itMSC - placebo vs. placebo - itMSC) as covariates.
  Participants
    Class II | 21
    Class III | 1
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 120 (17.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 74 (9.6)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 78 (14.2)
N-terminlal-proB-type Natriuretic Peptide (NT-proBNP) [Mean (Standard Deviation); unit: pg/mL] | 212 (841)
Troponin I [Mean (Standard Deviation); unit: ug/mL] | 0.0009 (0.0003)
Serum Sodium [Mean (Standard Deviation); unit: mmol/L] | 138 (2)
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.96 (0.23)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: International Units/milliliter (IU/mL)] | 21.86 (8.64)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] | 21.82 (9.57)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.4)
Albumin [Mean (Standard Deviation); unit: g/dL] | 4.2 (0.36)
History of Hypertension [Count of Participants; unit: Participants] | 5
History of Diabetes [Count of Participants; unit: Participants] | 3
History of Atrial Fibrillation [Count of Participants; unit: Participants] | 2
History of Kidney Disease [Count of Participants; unit: Participants] | 1
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 31.6 (9.8)
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: mL] | 189.6 (114.2)
Left Ventricular End-Diastolic Volume (LVEDV) [Mean (Standard Deviation); unit: mL] | 264.9 (120.4)
Loop diuretic medication [Count of Participants; unit: Participants] | 16
angiotensin converting enzyme inhibitors (ACEI) or Angiotensin II Receptor Blockers (ARB) medication [Count of Participants; unit: Participants] | 22
Mineralocorticoid Receptor Antagonist medication [Count of Participants; unit: Participants] | 18
Beta-blocker [Count of Participants; unit: Participants] | 22

OUTCOME MEASURES:

1. Primary Outcome: Safety Will be Evaluated by Number of AE
Description: As identified in the SAP, the safety analysis was the primary objective and was evaluated by the number of AEs
Time Frame: Total AEs and SAEs within 450 days post-infusion
Population: All 22 participants that received itMSC treatment were included. All adverse events are divided into serious and non-serious.
Measure: Number; unit: number of events
Groups:
- Experimental: Participants received itMSC
- Placebo: Participants received Placebo
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 22 | 20
number of events
  Adverse Events | 38 | 35
  Serious Adverse Events | 1 | 1
  Cell related adverse events | 1 | 0
  All-cause hospitalization | 0 | 0
  All-cause death | 0 | 0

2. Secondary Outcome: Change in LVEF From Baseline to Day 90 Post-initial Infusion.
Description: The secondary efficacy endpoint was the change in LVEF from baseline to Day 90 post-initial infusion. Participants with data available at each time point.
Time Frame: Baseline to Day 90
Population: The secondary efficacy endpoint according to the protocol was the change in LVEF from baseline to Day 90 post-initial infusion.
Measure: Mean (Standard Deviation); unit: percentage of ejection volume
Groups:
- Experimental: Human (itMSC): Intervention: One time intravenous infusion of 1.5 million (aMBMC) per kg administered at approximately 2mL/min. Maximum dose as for 100kg subject or 150 million cells for any subject 100kg or more.
  Allogeneic Mesenchymal Bone Marrow Cells (itMSC): One time infusion Allogeneic Mesenchymal Bone Marrow Cells (itMSC) 1.5 million cells/kg.
Arm/Group | Experimental: Human (itMSC) | Placebo:Lactated Ringer's Solution (LRS)
Number analyzed (Participants) | 12 | 12
percentage of ejection volume
  Baseline (%) | 34.3 (7.91) | 34.5 (7.49)
  90 days (%): number analyzed (Participants) | 9 | 12
  90 days (%) | 34.1 (9.7) | 36.7 (5.42)

ADVERSE EVENTS:
Time Frame: 450 days
Description: All AE summaries were restricted to treatment-emergent adverse events (TEAEs), and TEAEs were defined as those AEs with onset after the first dose of study treatment or existing events that worsened after the first dose during the study.
  Treatment-emergent AEs by severity (severe, other), relationship to study treatment ("related" or "not related"). Reported treshold 5%.
Groups:
- Experimental: Subjects that received experimental drug, 22 subjects
- Placebo: Subjects that received placebo, 20 subjects
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/20
Other Adverse Events (participants affected / at risk) | 18/22 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=22) | Placebo (N=20)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=22) | Placebo (N=20)
General Disorders and administration site condition: chest pain, fatigue, pyrexia (General disorders) | 3 | 11
Venous Pressure Jugular Increased (Investigations) | 6 | 4
Upper Respiratory Tract, Nasopharyngitis (Infections and infestations) | 3 | 9
Fluid Overload, Dehydration (Metabolism and nutrition disorders) | 8 | 4
Dizziness, headache (Nervous system disorders) | 10 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT02467387/Prot_SAP_000.pdf